CLINICAL TRIAL: NCT00030303
Title: A Feasibility And Toxicity Study Of Vaccination With HSP70 For The Treatment Of Chronic Myelogenous Leukemia In Chronic Phase
Brief Title: Vaccine Therapy in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCHC-01117; CDR0000069127 (Registry Identifier: PDQ (Physician Data Query)); UCHC-7659; NCI-V01-1685
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — HSP70 Heat-Shock Proteins

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- vaccine (Experimental): recombinant 70-kD heat-shock protein
  Interventions: Biological: recombinant 70-kD heat-shock protein

INTERVENTIONS:
Biological: recombinant 70-kD heat-shock protein

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells may make the body build an immune response to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of vaccination with autologous heat shock protein 70 in patients with chronic phase chronic myelogenous leukemia.
* Determine the toxicity of this vaccination in these patients.

OUTLINE: Patients undergo leukapheresis to obtain peripheral mononuclear cells (PMNCs). Heat shock protein 70 (HSP70) is derived from the autologous PMNCs. Patients receive HSP70 intradermally once weekly for 8 weeks.

Patients are followed for 2 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic phase chronic myelogenous leukemia

  * Philadelphia chromosome positive
* Peripheral blast count no greater than 10%
* No molecular remission
* Less than 3 years since initial diagnosis
* No anticipation of requirement for bone marrow or stem cell transplantation for 6 months

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 10 g/dL
* Platelet count at least 20,000/mm^3

Hepatic:

* Bilirubin less than 2.0 times upper limit of normal (ULN)
* Transaminase less than 2.0 times ULN

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant active infection requiring hospitalization
* No other serious illness or significant behavioral or psychological problem that would preclude study involvement

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* Prior interferon alfa allowed
* No concurrent interferon alfa

Chemotherapy:

* Prior cytarabine or other cytotoxic agents allowed
* No concurrent cytarabine or other cytotoxic agents
* Concurrent hydroxyurea allowed

Endocrine therapy:

* No concurrent corticosteroid therapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent immunosuppressive medications
* Concurrent imatinib mesylate allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-01 (Actual); Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zihai Li, MD, PhD, Study Chair — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Result] Li Z, Qiao Y, Liu B, Laska EJ, Chakravarthi P, Kulko JM, Bona RD, Fang M, Hegde U, Moyo V, Tannenbaum SH, Menoret A, Gaffney J, Glynn L, Runowicz CD, Srivastava PK. Combination of imatinib mesylate with autologous leukocyte-derived heat shock protein and chronic myelogenous leukemia. Clin Cancer Res. 2005 Jun 15;11(12):4460-8. doi: 10.1158/1078-0432.CCR-05-0250. PMID 15958631